CLINICAL TRIAL: NCT04558073
Title: Prevention of Eating Disorders in At-Risk Female Students: Adaptation and Evaluation of Two Interventions in French-Speaking Switzerland
Brief Title: Evaluation of Two Eating Disorders Prevention Interventions in At-Risk Female Students With Body Dissatisfaction
Acronym: HEIDI-BP-HW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 99021
Record Dates: First submitted 2020-09-04; First posted 2020-09-22 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Body Dissatisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The participants and the collaborators performing the interventions will not be blinded to the conditions. In order to minimize bias, the main statistical analyses aimed at evaluating the hypotheses will be performed by a statistician blinded to the participants' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Body Project (BP) (Experimental): The BP intervention includes four one-hour sessions given over a month by two facilitators. The sessions will be held on a collaborative platform in groups of six people.
  Interventions: Behavioral: Body Project (BP)
- Healthy Weight Program (HW) (Experimental): The HW intervention includes four one-hour sessions given over a month by two facilitators. The sessions will be held on a collaborative platform in groups of six people.
  Interventions: Behavioral: Healthy Weight Program (HW)
- Waiting-list (WL) (No Intervention): The waiting list will consist of two assessments each separated by a one-month interval. Following this waiting time, participants will receive the BP intervention.

INTERVENTIONS:
Behavioral: Body Project (BP) — The BP intervention offers discussions and exercises to make participants realize the cost of pursuing social ideals valuing thinness. This produces "cognitive dissonance", a cognitive discomfort due to a contradiction between speech and beliefs, which motivates to modify one's beliefs. The curriculum includes discussions on techniques of the advertising industry and the unique ideal of beauty promoted worldwide, as well as on the costs of pursuing the thin-ideal. Participants are also challenged to try behaviours they avoid because their appearance bother them. Societal activism actions are also discussed.
  Arms: Body Project (BP)
Behavioral: Healthy Weight Program (HW) — The HW intervention allows participants to make personalized changes in their diet and physical activity each week gradually, to aim for a health-ideal rather than a thin-ideal. The intervention is based on small changes, based on behavioural change techniques. Advice is given on what types of changes introduce to promote health, and how to implement changes sustainably. Difficulties are discussed in the group with a problem-solving approach. The last session introduces a long-term view of lifestyle change.
  Arms: Healthy Weight Program (HW)

SUMMARY:
Eating disorders are psychopathologies with serious repercussions on the somatic, psychological and social level. Currently available treatments are unfortunately for now not fully efficient, therefore researchers have recommended to develop prevention initiatives. Until now, no study has been carried out in Switzerland to evaluate the efficacy of an intervention for the prevention of eating disorders.

The goal of the present study is to evaluate two eating disorders prevention intervention that have been largely validated in the US, called the Body Project (BP) and the Healthy Weight Program (HW). Both interventions target body dissatisfaction, which is a well-identified risk factor of eating disorders. They will be compared to a one-month waiting list. Because of the pandemic situation due to the Severe Acute Respiratory Syndrome coronavirus (COVID-19), both interventions will be delivered virtually via a collaborative platform. The sessions will be recorded to carry out a quality control.

To compare the BP and HW interventions to a waiting list, a three-arm randomized controlled study will be carried out, including female students from French-speaking Switzerland. Recruitment will include 90 participants. Participants will be randomly assigned to one of the three arms of the study. They will be evaluated before (T0) and after (T1) the interventions or the waiting list. Following the interventions, the participants will have one month of follow-up before a final evaluation (T2). Participants on the waiting list will receive the BP following the one-month waiting period and will then be evaluated (T2).

After having signed the consent form, the participant will be randomized to one of the three study arms, with a 1: 1: 1 allocation ratio. Interventions will be given in groups of six participants. Randomization will be blocked to ensure groups of equal size, and that groups of six participants for each arm are regularly formed. The blocks will be of variable size (3, 6, 9) to protect the concealment.

The hypotheses are as follows:

1. The two interventions BP and HW will have an effect on body dissatisfaction (primary outcome) as well as on the thin-ideal internalization, dietary restraint, negative affect, and eating disorders psychopathology (secondary outcomes), compared to the waiting list;
2. There will be no differences between the BP and the HW on the primary and secondary outcomes;
3. The effects observed thanks to the interventions will be maintained after one month of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female student;
* Aged between 18 and 25 years old;
* BMI between 18.5 and 30 kg/m2;
* French-speaking (or understand French sufficiently to participate in the intervention) and having lived in Switzerland for at least six months;
* Suffering from body dissatisfaction and obtain a score of at least 26 on the Body Shape Questionnaire 8-item (BSQ-8C) which represents a moderate concern with her body image;
* Accepting the use of a collaborative platform to participate in the intervention group, which implies that her name may be revealed, and accept that the sessions be recorded.

Exclusion Criteria:

* Eating disorder according to the Diagnostic and Statistical Manuel of Mental Disorders 5th edition (DSM-5) diagnostic criteria (past or current);
* Diagnosis of mood disorder or anxiety disorder;
* Pregnancy.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Mean Change in Body Dissatisfaction on the Body Shape Questionnaire 8C (score ranging from 8 to 48, with higher scores indicating higher body dissatisfaction) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in Body Dissatisfaction after interventions in comparison with waiting-list

SECONDARY OUTCOMES:
Mean Change in Thin-Ideal Internalization on the Socio-Cultural Attitudes Towards Appearance Questionnaire (score ranging from 1 to 5 with higher scores indicating higher thin-ideal internalization) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in thin-ideal internalization after interventions in comparison with waiting-list
Mean Change in Dietary Restraint on the Dutch Eating Behaviour Questionnaire (score ranging from 1 to 5 with higher scores indicating higher dietary restraint) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in Dietary Restraint after interventions in comparison with waiting-list
Mean Change in Anxiety on the Hospital Anxiety and Depression Scale (score ranging from 0 to 21 with higher scores indicating higher anxiety) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in Anxiety after interventions in comparison with waiting-list
Mean Change in Depression on the Hospital Anxiety and Depression Scale (score ranging from 0 to 21 with higher scores indicating higher depression) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in Depression after interventions in comparison with waiting-list
Mean Change in Eating Disorders Psychopathology on the Eating Disorders Examination-Questionnaire (score ranging from 0 to 6 with higher scores indicating higher eating disorders psychopathology) from baseline to post-intervention or post-waiting | one month (Month 1)
  Mean change in Eating Disorders Psychopathology after interventions in comparison with waiting-list
Mean Change in Body Dissatisfaction on the Body Shape Questionnaire 8C (score ranging from 8 to 48, with higher scores indicating higher body dissatisfaction) from post-intervention to follow-up | one month (Month 2)
  Mean change in Body Dissatisfaction between post-intervention and follow-up
Mean Change in Thin-Ideal Internalization on the Socio-Cultural Attitudes Towards Appearance Questionnaire (score ranging from 1 to 5 with higher scores indicating higher thin-ideal internalization) from post-intervention to follow-up | one month (Month 2)
  Mean change in Thin-Ideal Internalization between post-intervention and follow-up
Mean Change in Dietary Restraint on the Dutch Eating Behaviour Questionnaire (score ranging from 1 to 5 with higher scores indicating higher dietary restraint) from post-intervention to follow-up | one month (Month 2)
  Mean change in Dietary Restraint between post-intervention and follow-up
Mean Change in Anxiety on the Hospital Anxiety and Depression Scale (score ranging from 0 to 21 with higher scores indicating higher anxiety) from post-intervention to follow-up | one month (Month 2)
  Mean change in Anxiety between post-intervention and follow-up
Mean Change in Depression on the Hospital Anxiety and Depression Scale (score ranging from 0 to 21 with higher scores indicating higher depression) from post-intervention to follow-up | one month (Month 2)
  Mean change in Depression between post-intervention and follow-up
Mean Change in Eating Disorders Psychopathology on the Eating Disorders Examination-Questionnaire (score ranging from 0 to 6 with higher scores indicating higher eating disorders psychopathology) from post-intervention to follow-up | one month (Month 2)
  Mean change in Eating Disorders Psychopathology between post-intervention and follow-up

OTHER OUTCOMES:
Mean of four 5-point Likert scales assessing program usefullness, help, understandability, usefulness of exercises (score from 1 to 5 with 5 indicating higher satisfaction) after interventions | Month 1 or Month 2
  Mean of satisfaction with BP and HW assessed with four Likert scales after interventions

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Carrard, PhD, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- School of Health Sciences (HES-SO Geneva), Geneva, Carouge, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the data will be stored in a repository which guarantees archiving and data sharing in accordance with Findability, Accessibility, Interoperability, and Reuse of digital assets (FAIR) principles.

REFERENCES:
- [Derived] Carrard I, Cekic S, Bucher Della Torre S. A randomized controlled trial to evaluate the acceptability and effectiveness of two eating disorders prevention interventions: the HEIDI BP-HW project. BMC Womens Health. 2023 Aug 23;23(1):446. doi: 10.1186/s12905-023-02607-6. PMID 37612687